CLINICAL TRIAL: NCT05812105
Title: Improving the Mobility of Transportation Disadvantaged Older Adults A Community-Based Intervention for the Hispanic/Latino Population
Brief Title: Improving the Mobility of Transportation Disadvantaged Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: Center for Transportation, Equity, Decisions and Dollars (Unknown); University of South Florida (Other)
Responsible Party: Principal Investigator, Kathy Lee, Assistant Professor, The University of Texas at Arlington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0391
Record Dates: First submitted 2023-03-20; First posted 2023-04-13 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Lack of Resources; Lack of Mobility
Keywords: Community; Education; Minority; Mobility; Social support

STUDY DESIGN:
Intervention Model Description: Participants received an intervention (i.e., Healthy Buddy Program providing a list of transportation/aging/health-related services available in their community) and complete pre- and post-surveys & interviews.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Buddy Program (Experimental): This intergenerational program targets Spanish speaking older adults who lack reliable and/or safe transportation and are managing at least one chronic illness. The program goal is to improve older adults' awareness of existing community resources, with an emphasis on transportation and health assets. Trained college students acted as facilitators for the program and helped older adults with relevant community resources.
  Interventions: Other: Healthy Buddy Program

INTERVENTIONS:
Other: Healthy Buddy Program — The Healthy Buddy Program is a community-based initiative that pairs college students with transportation disadvantaged, community- dwelling older adults age 65 and older. The Spanish-language Healthy Buddy Program was developed to measure the transportation and health challenges of Hispanic/Latino older adults and determine the efficacy of the adapted HB program model.

SUMMARY:
The primary objective of the research was to improve mobility for transportation-disadvantaged older adults by expanding the scope of the existing Healthy Buddy Program, to accommodate an aging Spanish-speaking population in the U.S.

DETAILED DESCRIPTION:
The research identified barriers and opportunities to improve Hispanic/Latino older adult access to community-based transportation and health resources. It was conducted with the existing Healthy Buddy model, which pairs older adults with college students who are trained to help them identify relevant transportation and health resources, while accommodating the unique needs of this transportation-disadvantaged population. The research team reevaluated the potential effectiveness of a Spanish-language accessible Healthy Buddy program model for increasing the self-efficacy and quality of life among Hispanic/Latino older adults. The team recruited bilingual (English-Spanish-speaking) students from multidisciplinary backgrounds. Older adult participants were invited to participate in pre- and post-surveys, including a qualitative interview, to allow the team to further evaluate the success of the program among Hispanic/Latino participants and to determine the replicability of the project in other communities with a significant population of transportation disadvantaged Hispanic/Latino older adults.

ELIGIBILITY:
Inclusion Criteria:

* Older adults age 65+
* Those who no longer drive
* Resident of Texas
* Those who manage at least one health condition (e.g., diabetes, high blood pressure, etc.)
* Spanish is primary language

Exclusion Criteria:

* Those who do not have a capacity to answer the pre-screening questions due to their cognitive and physical limitations
* Hispanic individuals who can speak fluent English will be excluded because they may have a better understanding of existing resources and information written and serviced in English in the community.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Quality of life and well-being of older adults | 4 weeks
  The title of the scale is Brief Older People's Quality of Life questionnaire. It is the short, 13-item version of the original Older People's Quality of Life questionnaire. Each of the 13 items is scored Strongly agree=5, Agree=4, Neither=3, Disagree=2, Strongly disagree=1. The items are summed for a total score, so that higher scores represented higher quality of life. The score ranges from 13 to 65.

SECONDARY OUTCOMES:
Self-efficacy correlated to emotion, stress, and health complaints | 4 weeks
  The title of the scale is General Self-Efficacy scale. The General Self-Efficacy Scale has 10 items correlated to emotion, optimism, work satisfaction. Each item is scored Not at all true=1, Hardly true=2, Moderately true=3, and Exactly true=4. The total score is calculated by finding the sum of the all items.The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Arlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37). Windsor, UK: NFER-NELSON.
- [Background] Bowling A, Hankins M, Windle G, Bilotta C, Grant R. A short measure of quality of life in older age: the performance of the brief Older People's Quality of Life questionnaire (OPQOL-brief). Arch Gerontol Geriatr. 2013 Jan-Feb;56(1):181-7. doi: 10.1016/j.archger.2012.08.012. Epub 2012 Sep 19. PMID 22999305

DOCUMENTS (1):
  • Informed Consent Form (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT05812105/ICF_000.pdf